CLINICAL TRIAL: NCT02767544
Title: Vaginal Wound Infiltration Analgesia for Postoperative Pain After Laparoscopic Hysterectomy: a Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Päivi Päkarinen, MD PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 98/13/03/03/2014/2
Record Dates: First submitted 2016-05-02; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Pain
Keywords: laparoscopic hysterectomy; postoperative pain; local analgesia; vaginal wound
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropivacaine group (Experimental): Vaginal wound local analgesia by 10ml ropivacaine 7.5mg/ml injection after laparoscopic hysterectomy
  Interventions: Procedure: Vaginal wound local analgesia after laparoscopic hysterectomy
- Control group (No Intervention): Vaginal wound no local analgesia by 10 ml ropivacaine 7.5mg/ml injection after laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Vaginal wound local analgesia after laparoscopic hysterectomy
  Arms: ropivacaine group

SUMMARY:
In cases of laparoscopic hysterectomy , women were randomized to two groups: ropivacaine ( vaginal wound infiltration analgesia) vs. control group. Results regarding postoperative pain and need of oxycodone.

DETAILED DESCRIPTION:
Women assigned to laparoscopic hysterectomy were randomly divided into two groups as regard surgery: a ropivacaine group (RG) (n=41) and a control group (CG) (n=40). General anesthesia and use of local anesthetics were standardized. Visual analog scale (VAS) scores for pain and side effects (nausea/vomiting) and the amount of postoperative analgesic used were recorded for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

The criteria for inclusion were scheduled laparoscopic hysterectomy

Exclusion Criteria:

The exclusion Criteria were contraindications to any of the forms of medication used in the study (oxycodone, ketoprofen, paracetamol), language difficulties ( inability to understand and speak Finnish or Swedish)

Ages: 30 Years to 80 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain scores | Change in 24 hours after surgery
  Visual Analog Score (VAS) for pain. Physicians Global Assessment to measure quality of pain. 10-point VAS score for pain (0-10), 0 indicating no pain and 10 indicating unbearable pain at 1,3,6,12 and 24 h (hour) after surgery (Units on a Scale; 0-10).

SECONDARY OUTCOMES:
Complication | Up to one week
  Frequency of complications. Values are given as n (%) and eventual complications are specified.
Nausea | Change in 24 hours after surgery.
  Nausea after the procedure: Visual Analog Score (VAS) for nausea. Physicians Global Assessment to measure quality of nausea. 10-point VAS score for nausea (0-10), 0 indicating no nausea and 10 indicating unbearable nausea at 1,3,6,12 and 24 h (hour) after surgery. ( Unit on scale; 0-10).
Length of hospitalisation | Up to one week
  Length of hospital stay measured from the end of the operation until discharge
The use of analgesics for postoperative pain | Change in 24 hours after surgery
  Postoperative pain defined by the total amount of analgesics used. Amount of used Oxycodone (mg).
Vomiting | Change in 24 hours after surgery.
  Vomiting after the procedure: Visual Analog Score (VAS) for vomiting. Physicians Global Assessment to measure quality of vomiting. 10-point VAS score for vomiting (0-10), 0 indicating no vomiting and 10 indicating unbearable vomiting at 1,3,6,12 and 24 h (hour) after surgery. ( Unit on scale; 0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Päivi I Pakarinen, MD PhD, Principal Investigator — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. A randomized controlled trial of perioperative administration of pregabalin for pain after laparoscopic hysterectomy. Pain. 2008 Jan;134(1-2):106-12. doi: 10.1016/j.pain.2007.04.002. Epub 2007 May 15. PMID 17507163
- [Background] Brummer TH, Jalkanen J, Fraser J, Heikkinen AM, Kauko M, Makinen J, Puistola U, Sjoberg J, Tomas E, Harkki P. FINHYST 2006--national prospective 1-year survey of 5,279 hysterectomies. Hum Reprod. 2009 Oct;24(10):2515-22. doi: 10.1093/humrep/dep229. Epub 2009 Jul 10. PMID 19592483
- [Background] Hristovska AM, Kristensen BB, Rasmussen MA, Rasmussen YH, Elving LB, Nielsen CV, Kehlet H. Effect of systematic local infiltration analgesia on postoperative pain in vaginal hysterectomy: a randomized, placebo-controlled trial. Acta Obstet Gynecol Scand. 2014 Mar;93(3):233-8. doi: 10.1111/aogs.12319. PMID 24576202
- [Background] Beaussier M, Bouaziz H, Aubrun F, Belbachir A, Binhas M, Bloc S, Fuzier R, Jochum D, Nouette-Gaulain K, Paqueron X; membres du comite douleur-ALR de Sfar. [Wound infiltration with local anesthetics for postoperative analgesia. Results of a national survey about its practice in France]. Ann Fr Anesth Reanim. 2012 Feb;31(2):120-5. doi: 10.1016/j.annfar.2011.10.017. Epub 2011 Dec 29. French. PMID 22209702
- [Background] Kato J, Ogawa S, Katz J, Nagai H, Kashiwazaki M, Saeki H, Suzuki H. Effects of presurgical local infiltration of bupivacaine in the surgical field on postsurgical wound pain in laparoscopic gynecologic examinations: a possible preemptive analgesic effect. Clin J Pain. 2000 Mar;16(1):12-7. doi: 10.1097/00002508-200003000-00003. PMID 10741813
- [Background] Kahokehr A, Sammour T, Srinivasa S, Hill AG. Systematic review and meta-analysis of intraperitoneal local anaesthetic for pain reduction after laparoscopic gastric procedures. Br J Surg. 2011 Jan;98(1):29-36. doi: 10.1002/bjs.7293. PMID 20979101